CLINICAL TRIAL: NCT04282720
Title: Hiatal Hernia Repair Using Surgimend Mesh: A Pilot Study
Brief Title: SurgiMend Mesh at the Hiatus
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kettering Health Network (Other)
Collaborators: Integra LifeSciences Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: SurgiMend
Record Dates: First submitted 2020-02-21; First posted 2020-02-25 (Actual); Last update posted 2023-10-05 (Actual); Status verified 2023-03

CONDITIONS: Hiatal Hernia
MeSH Terms: conditions — Hernia, Hiatal

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- SurgiMend Mesh (Other): SurgiMend Mesh - FDA approved noncross-linked bovine dermis biologic mesh. SurgiMend Mesh will be used according to FDA approved recommendations for the use of abdominal wall hernia reinforcement.
  SurgiMend is intended for implantation to reinforce soft tissue where weakness exists and for surgical repair of damaged or ruptured soft tissue membranes. SurgiMend is specifically indicated for:
  Hernia repair including abdominal, inguinal, femoral, diaphragmatic, scrotal, umbilical, and incisional hernias.
  Interventions: Device: SurgiMend Mesh

INTERVENTIONS:
Device: SurgiMend Mesh — Following placement of SurgiMend mesh during laparoscopic hiatal hernia repair, patient will be scheduled for follow up using an upper GI series to check for recurrence of the hiatal hernia. Follow up upper GIs will be performed at 6 months post-surgery. Subjects will also complete a QOL survey to assess other GI associated symptoms before and after surgical repair. The QOL survey can be administered by phone by study team members

SUMMARY:
Prospective, single-arm, open-label study to evaluate re-occurrence and quality of life in subjects undergoing primary Hiatal hernia repair using SurgiMend biological mesh. Up to 15, with a target of 10, subjects are planned to be enrolled at one site. All subjects will receive the SurgiMend mesh during surgery. Data collected will be compared to historical data.

Subjects will complete a pre-operative visit. After surgery, in addition to any standard of care visits, subjects will complete 3- and 6-month follow-ups involving a phone QOL survey and will have an upper GI series at 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of type 3 or 4 hiatal hernia (8)
* Subject is able to give informed consent
* Adults at least 18 years of age

Exclusion Criteria:

* Currently pregnant
* Prior hiatal hernia repair
* Prior gastric surgery
* Prior foregut surgery
* Known esophageal dysfunction or dysmotility
* Cirrhosis or ascites
* Known malignancy
* Known allergy to biologic mesh
* Known allergy to barium or other contrast material used in UGI
* Religious objection to animal implant
* Cognitive impairment
* Prisoners

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2020-03-31 (Actual); Primary Completion 2023-08-16 (Actual); Study Completion 2023-09-05 (Actual)

PRIMARY OUTCOMES:
Recurrence Rate | 6 months post surgery
  Recurrence rate will be analyzed by a Upper gastrointestinal tract radiography (UGI) and clinical evaluation in conjunction with patient's reported physiological assessment per the GERD-HRQL.

SECONDARY OUTCOMES:
Quality of Life Using GERD-HRQL Scale | pre-operative and 3 month and 6 month post surgery
  The GERD-HRQL was initially developed to measure the typical symptoms of GERD and their effect on a patient's quality of life. It was initially determined to have face validity and subsequent studies assessed its content validity and criterion validity. Reliability was determined by the test-retest method. This instrument is practical, with little administrative burden and has been validated for use via the telephone call. Scale is 0-5 with 0 being no symptoms and 5 being symptoms are incapacitating.

CONTACTS AND LOCATIONS:
Overall Officials: Paul Levy, DO, Principal Investigator — Kettering Health Network
Locations (1):
- Kettering Health Network - Grandview Medical Center, Dayton, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Furnee E, Hazebroek E. Mesh in laparoscopic large hiatal hernia repair: a systematic review of the literature. Surg Endosc. 2013 Nov;27(11):3998-4008. doi: 10.1007/s00464-013-3036-y. Epub 2013 Jun 21. PMID 23793804
- [Background] Lidor AO, Steele KE, Stem M, Fleming RM, Schweitzer MA, Marohn MR. Long-term quality of life and risk factors for recurrence after laparoscopic repair of paraesophageal hernia. JAMA Surg. 2015 May;150(5):424-31. doi: 10.1001/jamasurg.2015.25. PMID 25785415
- [Background] Nason KS, Luketich JD, Qureshi I, Keeley S, Trainor S, Awais O, Shende M, Landreneau RJ, Jobe BA, Pennathur A. Laparoscopic repair of giant paraesophageal hernia results in long-term patient satisfaction and a durable repair. J Gastrointest Surg. 2008 Dec;12(12):2066-75; discussion 2075-7. doi: 10.1007/s11605-008-0712-7. Epub 2008 Oct 8. PMID 18841422
- [Background] Adelman DM, Selber JC, Butler CE. Bovine versus Porcine Acellular Dermal Matrix: A Comparison of Mechanical Properties. Plast Reconstr Surg Glob Open. 2014 Jun 6;2(5):e155. doi: 10.1097/GOX.0000000000000072. eCollection 2014 May. PMID 25289348
- [Background] Velanovich V. The development of the GERD-HRQL symptom severity instrument. Dis Esophagus. 2007;20(2):130-4. doi: 10.1111/j.1442-2050.2007.00658.x. PMID 17439596
- [Background] Radiologic Society of North America (2019). Radiation dose in X-Ray and CT Exam. Available at https://www.radiologyinfo.org/en/info.cfm?pg=safety-xray
- [Background] K. S. Silvipriya, K. Krishna Kumar*, A. R. Bhat, B. Dinesh Kumar, Anish John, Panayappan Lakshmanan. Collagen: Animal Sources and Biomedical Application. Journal of Applied Pharmaceutical Science Vol. 5 (03), pp. 123-127, March, 2015. DOI: 10.7324/JAPS.2015.50322
- [Background] Kahrilas PJ, Kim HC, Pandolfino JE. Approaches to the diagnosis and grading of hiatal hernia. Best Pract Res Clin Gastroenterol. 2008;22(4):601-16. doi: 10.1016/j.bpg.2007.12.007. PMID 18656819